CLINICAL TRIAL: NCT01586832
Title: Stocking of a Busy Emergency Department
Status: Completed | Type: Observational
Sponsor: Lehigh Valley Hospital (Other)
Responsible Party: Principal Investigator, Marna Rayl Greenberg, Director of Emergency Medicine Research, Lehigh Valley Hospital
Other Study IDs: 2-20080104
Record Dates: First submitted 2011-07-19; First posted 2012-04-27 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Emergencies
Keywords: Hospital Supplies; Stocking of Supplies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ED Nurses: Nurses in the emergency department (ED) providing patient care using supplies found in the "stocking towers"

SUMMARY:
Stocking of essential supplies in an emergency department (ED) is crucial in order to efficiently and effectively take care of patients. When equipment and supplies are not available to patient care providers, an imbalance in the delivery of care is created. The amount of time nurses spend away from the bedside obtaining supplies has only been superficially studied; however, one study proposed that the majority of nurses spend 5 to 20 percent or more of their time during a shift. This results in 30 minutes to two-and-a-half hours of a twelve hour shift being lost to retrieving supplies that are not available.

Cabinets and drawers have recently been eliminated in the rooms and stock is kept in "supply towers" that contain all the necessary supplies to adequately take care of patients with the exception of medications, or stationary supplies. Towers are restocked every morning by a stocking technician by taking the towers to the stock room, resupplying them based on previously established PAR levels, and utilizing a standard chart that describes exactly what supply, and how many to stock within a specified area of the cart.

During their shift, the stocking technician must also respond to pages concerning low stock levels.

Hypothesis:

Nurses spend a significant amount of time away from the patient bedside during their shift looking for supplies.

DETAILED DESCRIPTION:
Objectives:

* Determine the amount of time nurses spend outside of a patient room obtaining supplies to care for the patient.
* Determine what supplies are obtained when the room is left.
* Determine how many times per shift the nurse leaves to obtain the same item.
* Determine if utilizing a "supply tower" located in patient rooms decreases the amount of time nurses spend obtaining supplies outside of a patient room to care for patients.
* Determine if implementation of a full time stocking technician decreases the amount of time that nurses spend outside a patient's room obtaining stock.
* Conduct spot checks on carts to determine if PAR levels are over, under, or exactly as established.

ELIGIBILITY:
Inclusion Criteria:

* Nurse is an employee of LVHHN, and is working at the CC site.
* Nurse is working a full shift (7a-7p, 7p-7a, 7a-3p, 3p-11p, 11p-7a).
* The nurse being observed is working in Pod 1, Pod 2, Pod 3, or Pod 4 at the CC site.
* The supply needed is related to a procedural task for patient care.

Exclusion Criteria:

* The nurse is working at LVH-M or LVH-17.
* The nurse being observed is working in the express care area or trauma bay.
* The supply being obtained is a supply that is not maintained in the cart (Appendix 2).
* The nurse is scheduled for a shift less than 8 hours.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will include the nurses in the emergency department who will be observed during their shift.
Sampling Method: Non-Probability Sample
Enrollment: 565 (Actual)
Dates: Start 2008-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
time nurses spend away from patients bedside | Outcome will be assessed for one year as the average time nurses spend away from the bedside searching for supplies for patient care during an ED stay (an expected average of 2.5 hours)
  The average time nurses spend away from the bedside searching for supplies for patient care during an ED stay (an expected average of 2.5 hours)

SECONDARY OUTCOMES:
Supplies searched for | Outcome will be assessed for one year as the type of supply that the nurses are searching for that was not available at the bedside searching for supplies for patient care during an ED stay (an expected average of 2.5 hours)
  This is the type of supply that the nurse was searching for that was not available at the bedside.

CONTACTS AND LOCATIONS:
Overall Officials: David Richardson, MD, Principal Investigator — Lehigh Valley Health Network
Locations (1):
- Lehigh Valley Health Network, Allentown, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
However, the overall study results were published in JONA, vol 44, issue 11, November, 2014.